CLINICAL TRIAL: NCT01561495
Title: Proton Radiotherapy for Extremity Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Request- Global low enrollment
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 09510
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Soft Tissue Sarcoma of the Extremities
Keywords: scheduled to receive RT either pre- or postoperatively
MeSH Terms: interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Participants (Experimental): Proton Radiotherapy
  Interventions: Radiation: Proton Therapy

INTERVENTIONS:
Radiation: Proton Therapy

SUMMARY:
This is a study of proton radiotherapy for the pre- or post- operative treatment of patients with extremity sarcoma. This study will treat patients in two dose groups:

1. patients receiving pre-operative proton therapy and
2. patients receiving post-operative proton therapy. In each dose group, the study is divided into two phases. In the first phase of the study, the investigators will determine if treatment with proton therapy is safe and can be delivered on a regular basis. In the second phase, the investigators will determine if proton therapy has less long term side effects compared to standard radiation in both pre-operative patients and post-operative patients.

DETAILED DESCRIPTION:
This study will be performed in two phases. In the first phase, feasibility will be established using the primary objectives set below. The second part will begin no earlier than 30 days after the last patient in the initial phase has completed treatment and once safety and feasibility has been verified.

The primary objective of this study is feasibility. The study will be deemed infeasible if 10% or more of patients experience one of the following:

1. Patient cannot be given treatment because anatomy is such that a dosimetrically satisfactory treatment plan cannot be devised (95% of planning target volume covered by 95% of the dose).
2. Patient is unable to tolerate more than 25% of treatments (for any reasonable to set patient up within acceptable limits of tolerance, patient unable to tolerate treatment position or immobilization for duration of treatment) using proton radiotherapy. Note: this end-point is proton-therapy specific, and indicates feasibility of proton as opposed to photon radiotherapy. For example, if the proton-specific patient immobilization/positioning is not well tolerated or extra time in the treatment position is too long or uncomfortable, protons delivered per protocol would be deemed not feasible compared to photons. Any treatments that cannot be delivered with protons will be delivered using photons, so that the patient receives the prescribed tumor dose.
3. Patient is unable to complete all of his/her treatments within 10 days of estimated date of treatment completion or requires a treatment break greater than 5 days. Additionally, no greater than 33% of patients experience a significant toxicity.

Primary Objectives for second phase of study are:

* The primary objective of Phase II in the pre-operative group will be to evaluate the wound complication rate of pre-operative proton radiotherapy in patients with STS of the lower extremity.
* The primary objective of Phase II in the post-operative group will be to evaluate the functional outcome (e.g., fibrosis, joint stiffness, edema) at two years after post-operative proton radiotherapy in patients with STS of the lower extremity.

Secondary Objectives for both phases of study are:

* To assess the local control rate, progression-free survival and overall survival of proton radiotherapy for STS of the extremity.
* To determine the acute and late toxicities of proton radiotherapy to the extremities.
* To monitor for effects of proton treatment on tumor and normal tissues using radiographic imaging (both cohorts) or ex-vivo analysis of tissue samples (pre-operative cohort only).
* To examine the relationship between pre-treatment hypoxia as determined by F18-EF5 scanning and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of soft tissue sarcoma of the extremities are eligible for this study.
* Patient must be 18 years of age.
* Patients must have evidence of disease limited to the extremities.
* For the pre-operative group, patients must be considered operable/resectable and a candidate for pre-operative radiotherapy as judged by the attending surgeon and radiation oncologist. The clinical evaluation of patients will include a work up as per the standard of care. All patients in the pre-operative group will be evaluated for this protocol PRIOR to the initiation of therapy.
* For the post-operative group, patients must be considered operable/resectable (if evaluated prior to resection) and a candidate for post-operative radiotherapy by the attending surgeon and radiation oncologist. The clinical evaluation of patients will include a work up as per the standard of care. Patients in the post-operative group may be evaluated PRIOR to the initiation of any therapy or may be referred for evaluation after surgical resection.
* ECOG status of 0-2.
* Patients must sign a document that indicates that they are aware of the investigative nature of the treatment of this protocol, and the potential benefits and risks. Patients unwilling or unable to sign informed consent are excluded from the study.
* Women of child-bearing potential as long as she agrees to use a recognized method of birth control (e.g. oral contraceptive, IUD, condoms or other barrier methods etc.). Hysterectomy or menopause must be clinically documented.
* Negative urine pregnancy test for females of childbearing potential on the day of the F18-EF5 PET scan prior to F18-EF5 injection

Exclusion Criteria:

* Pregnant women, women planning to become pregnant and women that are nursing.
* Patients who experience surgical complications that prevent radiation from starting for 5 months or more, unless there is evidence of gross residual disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06; Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtiland Deville, MD, Principal Investigator — Johns Hopkins Kimmel Cancer Center at Sibley Memorial Hospital
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All study participants received proton radiotherapy.
Period: Overall Study
Arm/Group | All Study Participants
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only one participant was enrolled.
Arm/Group | All Study Participants
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Given this is initially a feasibility study- the primary measure is number of AEs (Adverse Events).
Time Frame: 4 years
Population: Investigator and study team are unreachable after having left Penn despite multiple efforts to contact for more information- as such no data is available to present
Groups:
- All Participants: Proton Radiotherapy
  Proton Therapy
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years
Description: Investigator and study team are unreachable after having left Penn despite multiple efforts to contact for more information- as such no data is available to present. All information regarding Adverse Events are not accessible here at Penn.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-03-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT01561495/Prot_SAP_000.pdf
  • Informed Consent Form (2013-10-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT01561495/ICF_001.pdf